CLINICAL TRIAL: NCT02568930
Title: SUSTAIN-IT: Sustaining Quality of Life of the Aged: Heart Transplant or Mechanical Support?
Acronym: SUSTAIN-IT
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kathleen Grady, Professor, Feinberg School of Medicine, Northwestern University
Other Study IDs: STU00200851; 1R01AG047416 (NIH)
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
Keywords: quality of life heart failure mechanical support transplant
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Heart Transplantation (HT): The cohort includes advanced heart failure patients (60-80 years of age) listed for HT and their caregivers.
- Mechanical Circulatory Support (MCS): The cohort includes advanced heart failure patients (60-80 years of age) scheduled for DT MCS and their caregivers.

SUMMARY:
The purpose of this study is to compare health-related quality of life (HRQOL) outcomes in older (60-80 years) advanced heart failure (HF) patients who undergo heart transplantation (HT) or mechanical circulatory support (MCS) as a permanent implant (i.e., destination therapy [DT]) and their caregivers. Our study will contribute to better patient-centered care of older advanced HF patients and their caregivers, by informing decision making and guiding strategies to enhance post-operative HRQOL.

DETAILED DESCRIPTION:
The purpose of this study is to compare health-related quality of life (HRQOL) outcomes in older (60-80 years) advanced heart failure (HF) patients who undergo heart transplantation (HT) or mechanical circulatory support (MCS) as a permanent implant (i.e., destination therapy [DT]) and their caregivers, risk factors for poor HRQOL, adverse event and symptom burden, and quality-adjusted life years (QALYs). Advanced HF patients, 60-80 years of age, are an appropriate target group for this study because they are receiving HTs and MCS devices more frequently, and despite a greater risk for poor clinical outcomes, they have acceptable rates of survival. Using a prospective, longitudinal design, our multi-site comparative effectiveness research will compare HRQOL outcomes in patients who receive HT or DT MCS and their caregivers, from baseline to 2 years post-operatively. The primary aim of this proposed study is to determine whether older advanced HF patients who undergo DT MCS, as compared to patients who undergo HT, experience non-inferior change in overall HRQOL (primary), and domains of HRQOL (physical, mental, and social) from baseline through 2 years after surgery. Secondary Aims are (1.) to determine whether caregivers of older advanced HF patients who undergo DT MCS, compared to caregivers of older advanced HF patients who undergo HT, experience non-inferior change in overall HRQOL and domains from baseline through 2 years after surgery; (2.-3.) to identify risk factors related to poorer overall HRQOL in older DT MCS patients and their caregivers, as compared to older HT patients and their caregivers, at 2 years after surgery; (4.) to determine whether older advanced HF patients who undergo DT MCS, as compared to patients who undergo HT, have non-inferior rates of freedom from adverse events & symptoms at 1 and 2 years after surgery; and (5) to evaluate the distribution of QALYs in older advanced HF patients who undergo DT MCS, as compared to patients who undergo HT at 2 years after surgery. Our proposed study will contribute to better patient-centered care of older advanced HF patients and their caregivers, by informing decision making and guiding strategies to enhance post-operative HRQOL.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Advanced HF and listed with the United Network for Organ Sharing (UNOS) for a "primary" HT or scheduled to receive a "primary" DT LVAD;
2. Ages 60-80 years and able to speak, read, and understand English;
3. Willing to participate and ability to provide informed consent.

Caregiver Inclusion criteria:

1. Primary caregiver, identified by the patient, prior to DT MCS or while a candidate for HT;
2. Unpaid family member or friend who helps the patient with self-care;
3. Age > 21 years and able to speak, read, and write English;
4. Willing to participate and ability to provide informed consent.

Patient Exclusion criteria

1. Patient has a prior HT or MCS device
2. Patient is listed for multiple organ transplantation (i.e., heart/lung, heart/kidney, etc.)

Caregiver Exclusion criterion:

1) Patient refusal to participate.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes advanced heart failure patients (60-80 years of age) scheduled for DT MCS and their caregivers and advanced heart failure patients (60-80 years of age) listed for HT and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 694 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Non-inferior change in patient HRQOL | baseline through 2 years after surgery
  To determine whether older advanced HF patients who undergo DT MCS, as compared to patients who undergo HT, experience non-inferior change in overall HRQOL (primary outcome) and HRQOL domains (physical, mental, and social [secondary outcomes]) from baseline through 2 years after surgery.

SECONDARY OUTCOMES:
Non-inferior change in caregiver HRQOL | baseline through 2 years after surgery
  To determine whether caregivers of older advanced HF patients who undergo DT MCS, as compared to caregivers of older advanced HF patients who undergo HT, experience non-inferior change in overall HRQOL and HRQOL domains from baseline through 2 years after surgery.
Risk factors related to poorer patient overall HRQOL | 2 years after surgery
  To identify risk factors related to poorer overall HRQOL in older DT MCS patients, as compared to older HT patients, at 2 years after surgery.
Risk factors related to poorer caregiver overall HRQOL | 2 years after surgery
  To identify risk factors related to poorer overall HRQOL in caregivers of older DT MCS patients, as compared to caregivers of older HT patients, at 2 years after surgery.
Non-inferior rates of freedom from adverse events & symptoms | 1 and 2 years after surgery
  To determine whether older advanced HF patients who undergo DT MCS, as compared to patients who undergo HT, have non-inferior rates of freedom from adverse events & symptoms at 1 & 2 years after surgery.
Distribution of QALYs | 2 years after surgery
  To evaluate the distribution of QALYs in older advanced HF patients who undergo DT MCS, as compared to patients who undergo HT at 2 years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Grady, RN, PhD, Principal Investigator — Northwestern University
Locations (13):
- United States (13):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Florida Hospital, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Medical Center-Fairview Health Services, Minneapolis, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University (OSU), Columbus, Ohio
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Nguyen DD, Spertus JA, Benton MC, Thomas M, Jones PG, Andrei AC, Wu T, Baldridge AS, Grady KL. Association of Patient Reported Outcomes With Caregiver Burden in Older Patients With Advanced Heart Failure: Insights From the SUSTAIN-IT Study. Circ Heart Fail. 2024 Jul;17(7):e011705. doi: 10.1161/CIRCHEARTFAILURE.124.011705. Epub 2024 Jun 24. PMID 38910557
- [Derived] Chuzi S, Wilcox JE, Kao A, Spertus JA, Hsich E, Dew MA, Yancy CW, Pham DT, Hartupee J, Petty M, Cotts W, Pamboukian SV, Pagani FD, Lampert B, Johnson M, Murray M, Takeda K, Yuzefpolskaya M, Silvestry S, Kirklin JK, Wu T, Andrei AC, Baldridge A, Grady KL. Change in Caregiver Health-Related Quality of Life From Before to Early After Surgery: SUSTAIN-IT Study. Circ Heart Fail. 2023 Aug;16(8):e010038. doi: 10.1161/CIRCHEARTFAILURE.122.010038. Epub 2023 Jun 22. PMID 37345518
- [Derived] Okwuosa IS, Anderson A, Petty M, Wu T, Andrei AC, Kao A, Spertus JA, Pham DT, Yancy CW, Dew MA, Hsich E, Cotts W, Hartupee J, Pamboukian S, Pagani F, Lampert B, Johnson M, Murray M, Tekeda K, Yuzefpolskaya M, Kirklin JK, Grady KL. Caregiver burden before heart transplantation and long-term mechanical circulatory support: Findings from the sustaining quality of life of the aged: Transplant or mechanical support (SUSTAIN-IT) study. J Heart Lung Transplant. 2023 Sep;42(9):1197-1204. doi: 10.1016/j.healun.2023.01.015. Epub 2023 Apr 21. PMID 37088337
- [Derived] Grady KL, Kao A, Spertus JA, Hsich E, Dew MA, Pham DT, Hartupee J, Petty M, Cotts W, Pamboukian SV, Pagani FD, Lampert B, Johnson M, Murray M, Takeda K, Yuzefpolskaya M, Silvestry S, Kirklin JK, Andrei AC, Elenbaas C, Baldridge A, Yancy C. Health-Related Quality of Life in Older Patients With Heart Failure From Before to Early After Advanced Surgical Therapies: Findings From the SUSTAIN-IT Study. Circ Heart Fail. 2022 Oct;15(10):e009579. doi: 10.1161/CIRCHEARTFAILURE.122.009579. Epub 2022 Oct 10. PMID 36214123
- [Derived] Grady KL, Andrei AC, Elenbaas C, Warzecha A, Baldridge A, Kao A, Spertus JA, Pham DT, Dew MA, Hsich E, Cotts W, Hartupee J, Pamboukian SV, Pagani FD, Petty M, Lampert B, Johnson M, Murray M, Takeda K, Yuzefpolskaya M, Silvestry S, Kirklin JK, Yancy C. Health-Related Quality of Life in Older Patients With Advanced Heart Failure: Findings From the SUSTAIN-IT Study. J Am Heart Assoc. 2022 Feb 15;11(4):e024385. doi: 10.1161/JAHA.121.024385. Epub 2022 Feb 12. PMID 35156421

DOCUMENTS (1):
  • Informed Consent Form (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT02568930/ICF_000.pdf